CLINICAL TRIAL: NCT05154526
Title: Comparison of the Efficiency of Manual Therapy and Exercise in People With Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tuğba Akgüller (Other)
Responsible Party: Sponsor-Investigator, Tuğba Akgüller, Lecturer, Istanbul Arel University
Organization: Istanbul Arel University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Istanbul University Cerrahpasa
Record Dates: First submitted 2021-11-13; First posted 2021-12-13 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Neck Pain; Mobility Limitation
Keywords: neck pain; mechanical neck pain; manual therapy; exercise
MeSH Terms: conditions — Neck Pain; Mobility Limitation; Motor Activity | interventions — Musculoskeletal Manipulations; Resistance Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise Group (Experimental): Exercise Program only
  Interventions: Other: Exercise Program
- Manual Therapy Group (Active Comparator): Manual Therapy only
  Interventions: Other: Manual Therapy
- Manual Therapy and Exercise Group (Active Comparator): Manual Therapy + exercise program
  Interventions: Other: Manual Therapy; Other: Exercise Program

INTERVENTIONS:
Other: Manual Therapy — Manual Therapy: High velocity-low amplitude technique
  Arms: Manual Therapy Group; Manual Therapy and Exercise Group
Other: Exercise Program — Exercise program
  Arms: Exercise Group; Manual Therapy and Exercise Group

SUMMARY:
Mechanical neck pain (MNP) is defined as neck pain that becomes evident with the posture of the cervical region, movement or palpation of the cervical region muscles, felt in the cervical, occipital or posterior scapular region without spreading to the upper extremity, and without any trauma or specific pathology underlying the complaints. Most of the MNP cases are due to muscular or paraspinal soft tissue problems and show improvement in the first 6 weeks with conservative treatment methods. Various manual therapy techniques and various exercises are reported to have positive effects on neck pain. However, the isolated effects of these techniques in people with MNP are not fully known. Therefore, the aim of this study is to determine the effects of two different treatment programs in which the manual therapy technique and the exercise program are applied in individuals with MNP. In addition, comparing the effect of the treatment program in which manual therapy and exercise program are applied together with the isolated effects of these techniques is another aim.

DETAILED DESCRIPTION:
Mechanical neck pain (MNP) is defined as neck pain that becomes evident with the posture of the cervical region, movement or palpation of the cervical region muscles, felt in the cervical, occipital or posterior scapular region without spreading to the upper extremity, and without any trauma or specific pathology underlying the complaints. MNP causes symptoms such as pain in the cervical region, increased sensitivity to pressure, decrease in active range of motion (ROM) of the cervical region, drowsiness, and dizziness. Most of the MNP cases are due to muscular or paraspinal soft tissue problems and show improvement in the first 6 weeks with conservative treatment methods. When the current treatment recommendations are examined according to the duration of neck pain accompanied by limitation of movement, an exercise program that includes thoracic region mobilization, cervical ROM exercises, and strengthening and stretching exercises for the scapulothoracic region and upper extremity muscles is recommended for acute neck pain. In addition, various manual therapy techniques can be applied to the cervical region.

In subacute neck pain, an exercise program is applied to increase the endurance of the neck and upper extremity muscles. During this period, various manual therapy methods can be applied to the thoracic and cervical region. In chronic neck pain, combined treatment applications including various exercises, mobilization and manipulation techniques, dry needling, laser and intermittent manual/mechanical traction are recommended. It is stated that the high-velocity low-amplitude technique, which is among the manual therapy techniques and used in many musculoskeletal problems, can increase the ROM, decrease the pain and improve the function.

Various manual therapy techniques and various exercises are reported to have positive effects on neck pain. However, the isolated effects of these techniques in people with MNP are not fully known. Therefore, the aim of this study is to determine the effects of two different treatment programs in which the manual therapy technique and the exercise program are applied in individuals with MNP. In addition, comparing the effect of the treatment program in which manual therapy and exercise program are applied together with the isolated effects of these techniques is another aim.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MNP
* Decrease in cervical region ROM
* Ability to adapt to verbal, written and visual instructions

Exclusion Criteria:

* Spine surgery history
* Neurological neck pain in the cervical region
* Presence of tumor in the cervical region
* Blood coagulation disorders
* Vertebrobasilar artery insufficiency
* Cervical region trauma history
* Communicative/mental problems that prevent participation in treatment
* Inflammatory rheumatological diseases affecting the cervical region
* Physiotherapy and rehabilitation treatments for neck pain in the last 3 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-04-19 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | 6 weeks
  The neck function of the patients will be evaluated with the Neck Disability Index. The disability levels of the participants due to neck pain will be evaluated with the 'Neck Disability Index' . This scale consists of 10 items including pain intensity, personal care, lifting, reading, headache, concentration, work, driving, sleep status and leisure activities. Each item was scored from 0 (no disability) to 5 (complete disability).
Pain intensity | 6 weeks
  Pain intensity of the patients at rest, during activity and at night was assessed using the Visual Analog Scale (VAS). In this evaluation, individuals were told that the number "0" on the 10 cm long horizontal line expresses "no pain", and the number "10" indicates "unbearable pain" and that individuals should mark their intensity of pain on this line.

SECONDARY OUTCOMES:
Range of Motion (ROM) | 6 weeks
  Active neck flexion-extension, right-left lateral flexion and right-left rotation ROM of the participants will be evaluated with cervical goniometer.
Pain Pressure Threshold (PPT) | 6 weeks l
  Participants' PPTs will be evaluated with a pressure algometer (Baseline Push-Pull Force Gauge®, Fabrication Enterprises, Inc.) that can measure pressure in kilograms and pounds, with a 1 cm diameter circular rubber tip attached to the piston of the pressure gauge
36-Item Short Form Survey (SF-36) | 6 weeks
  Patients' quality of life will be evaluated with SF-36. This scale is a general health questionnaire that evaluates the person's perception of quality of life in the last four weeks under 8 sub-headings and 36 items. The sub-headings it includes; physical functions, physical roles, pain, social functions, mental health, emotional roles, energy and general health perception.
Patient satisfaction level | At the end of 6-weeks
  Patient Satisfaction will be assessed with the Global Rating of Change (GRC) scale. The scale to be used consists of 5 points (-2: I am much worse. -1: I am worse, 0: I am the same, +1: I am better, +2: I am much better).

CONTACTS AND LOCATIONS:
Overall Officials: Yıldız Analay Akbaba, PhD, Study Director — Istabul University-Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Buyukcekmece, Turkey (Türkiye)